CLINICAL TRIAL: NCT00035126
Title: An Open-Label Phase IIa Trial Evaluating the Safety and Efficacy of EPO906 as Therapy in Patients With Advanced Breast Cancer
Brief Title: EPO906 Therapy in Patients With Advanced Breast Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CEPO906A2205
Record Dates: First submitted 2002-05-02; First posted 2002-05-03 (Estimated); Last update posted 2017-02-08 (Estimated); Status verified 2017-02

CONDITIONS: Breast Neoplasms
Keywords: breast; cancer; tumor; tumour; intravenous; epothilone; taxane; anthracycline
MeSH Terms: conditions — Breast Neoplasms; Neoplasms | interventions — epothilone B

ARMS (1):
- EPO906 (Experimental)
  Interventions: Drug: epothilone b

INTERVENTIONS:
Drug: epothilone b

SUMMARY:
This study will examine whether the investigational drug EPO906, given by intravenous infusion (IV directly into the vein), is effective in shrinking tumors and preventing the growth of cells that cause breast cancer.

ELIGIBILITY:
Inclusion Criteria:

The following patients may be eligible for this study:

* Histologically or cytologically documented evidence of disease with at least one measurable lesion;
* Life expectancy of greater than three (3) months;
* Patients who have had only one prior therapy for metastatic disease;
* Patients who have received prior treatment with hormonal agents or who have had prior treatment regimens of radiotherapy in addition to one or no previous chemotherapy regimens are eligible;
* Patients who have had no prior therapy for metastatic disease, but who have received a taxane and an anthracycline (single or combination therapy) as adjuvant treatment, are eligible. For patients who have had previous radiation therapy to the target lesion(s), the lesion(s) must since have demonstrated progression.

Exclusion Criteria:

The following patients are not eligible for this study:

* Bone-only disease;
* Symptomatic pleural effusions;
* Symptomatic CNS metastases or leptomeningeal involvement;
* Any peripheral neuropathy or unresolved diarrhea greater than Grade 1;
* Severe cardiac insufficiency;
* Patients taking Coumadin or other warfarin-containing agents with the exception of low dose Coumadin (1 mg or less) for the maintenance of in-dwelling lines or ports;
* History of another malignancy within 5 years prior to study entry except curatively treated non-melanoma ckin cancer or cervical cancer in situ;
* Active or suspected acute or chronic uncontrolled infection including abcesses or fistulae;
* HIV+ patients;
* Pregnant or lactating females;
* Patients who have had radiation, chemotherapy, or hormonal therapy within the last four (4) weeks excluding palliative radiotherapy to isolated peripheral bone metastases not being used as markers for efficacy;
* Patients taking Herceptin less than three (3) weeks prior to study start.

Ages: 18 Years to 85 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 46 (Actual)
Dates: Start 2002-01 (Actual); Primary Completion 2003-11 (Actual); Study Completion 2003-11 (Actual)

PRIMARY OUTCOMES:
Tumor response as assessed by radiologic techniques and/or physical examination based on Response Evaluation Criteria in Solid Tumors (RECIST) | Every 8 weeks

SECONDARY OUTCOMES:
Time to progression | until disease progression, death or date of last follow-up
Overall survival | date of death or last date patient was known to be alive
Duration of overall response | every 8 weeks as clinically needed
Safety of study drug | weekly for the first 8 weeks, then every other week
pharmacokinectics of study drug | every 8 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (2):
- United States (2):
  - Dartmouth Hitchcock Medical Center, Lebanon, New Hampshire
  - Cancer Institute of New Jersey (CINJ), New Brunswick, New Jersey